CLINICAL TRIAL: NCT02861833
Title: Identifying Coping Strategies of Patients With Cancerous Wound After a Specific Nursing Accompaniment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_3976 - 2215
Record Dates: First submitted 2016-08-03; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Cancerous Wounds

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with a cancerous wound: major patients followed in a cancer ward and holders of a cancerous wound.
  Interventions: Other: nursing support

INTERVENTIONS:
Other: nursing support — Determining the Variability of adaptation strategies and correlations with specific nursing management, individual and contextual characteristics of patients with cancerous wounds

SUMMARY:
This is a first care research focuses on the study of adaptation strategies implemented by cancerous wound patients. Today, advances in treatment generally increases the life expectancy of a patient with cancer. the patients thus live longer with their wound. How to live then? The literature review shows that there is research on adaptation strategies in cancer pathology and that different factors seem to interact with these strategies. However the investigators have not found written on the theme cancerous wound and adaptation strategies.

the investigators conducted a pilot study of this research in medical oncology, Prof. service Duffaud CHU Timone, which allowed us to highlight patient adherence and motivation centers contacted but also areas for improvement. Indeed, the investigators now were doing a study of adaptation strategies implemented by the patient time T of his life. However, adaptation is a process in constant motion, the investigators want to identify two different time patients coping strategies following a specific charge nurse taking.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient having at least a cancerous wound.
* Patient having read the information leaflet and has given its consent.
* Patient able to meet a French language questionnaire.

Exclusion Criteria:

* History or active psychiatric illness.
* Unable to give informed consent.
* Inability to comply with the protocol procedures for geographical, social or psychological.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: major patients followed in a cancer ward and holders of a cancerous wound.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Descriptive analysis of the main demographic, clinical, and psychological | one month
  Questionnaires for patients rely on the concept of Coping,It refers to the responses and reactions that an individual develops to control aversive situation.

SECONDARY OUTCOMES:
main clinical features | one month
  The questionnaires are based on the concept of the coping, the nursing model on adaptation strategies developed by Callista Roy.
main psychological characteristics | one month
  The questionnaires are based on the concept of the coping, the nursing model on adaptation strategies developed by Callista Roy.

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille Hôpital de Timone, Marseille, France